CLINICAL TRIAL: NCT05397041
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of BMB-101 in Fed and Fasted Adult Healthy Human Volunteers
Brief Title: A 3-Part Study to Evaluate the Safety, Tolerability, PK, and Food Effect of BMB-101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bright Minds Biosciences Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-BMB-101-101
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: SAD, FE, MAD, dose escalating
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMB-101 (Experimental): Participants receiving BMB-101 orally
  Interventions: Drug: BMB-101
- Placebo (Placebo Comparator): Participants receiving Matched Placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMB-101 — Participants will receive one of several different oral doses of BMB-101 once or twice daily
  Arms: BMB-101
Drug: Placebo — Matched Placebo
  Arms: Placebo

SUMMARY:
This study is designed as a single centre, double blind, placebo controlled, randomized, SAD/FE/MAD, safety, tolerance and PK study of BMB-101 in healthy adult subjects. The study will be conducted as a 3-part study.

DETAILED DESCRIPTION:
This study is designed as a 3-part study:

Part 1 is designed as single ascending dose (SAD) escalation study investigating 4 dose levels. Each cohort will consist of participants to be randomly assigned to receive a blinded oral dose of BMB-101 or placebo.

Part 2 is designed as a randomized, orally administered, single-dose, two-treatment (fed vs fasted), two-period, two-sequence crossover to assess the effects of a standard high-fat breakfast on PK of BMB-101.

Part 3 is designed as a multiple ascending dose (MAD) escalation study investigating up to 4 dose levels. Subjects will be randomized to receive double-blind treatment of BMB-101 or matching placebo twice daily for 7 days.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject must be aged between 18 and 55 years (both inclusive).
2. Healthy subjects with no clinically significant screening results.
3. Body mass index (BMI) 18.0 to 32.0 kg/m².
4. Males and non pregnant females willing to use contraceptives consistent with local regulations from screening through 3 months after the last dose of study medication.
5. Agree to frequent blood and urine sampling during the course of the study.
6. Agree to be confined in the study unit and follow study procedures.

Key Exclusion Criteria:

1. Subjects with unstable or severe illness as indicated on medical history, physical examination, or clinical laboratory, vital signs, and electrocardiograms (ECGs) evaluations, or in the opinion of the Investigator.
2. Subjects with reported history within past 6 months of, or current treatment for, any GI disease that may impact the absorption of an oral drug for example gastroesophageal reflux disorder, peptic ulcer disease, inflammatory bowel disease.
3. Subjects with a history of seizures other than febrile seizures as a child.
4. Subjects with history of or current glucose intolerance; or with history of gestational diabetes.
5. Subjects with lifetime history of suicidal behavior or with lifetime history of suicidal ideation as indicated by the Columbia-Suicide Severity Rating Scale (C-SSRS)
6. Subjects with any use of or intent to use any medications, including prescription, over-the-counter (OTC), herbal preparations, or vitamin/mineral supplementation, other than study medications, from 7 days prior to first dose through follow-up visit.
7. Female subjects with a positive pregnancy test at Screening or Day -1 or who are breastfeeding.
8. Subjects who have used more than 5 cigarettes, cigars, or nicotine-containing products per month within 6 months prior to first study dose, or plan to use them through completion of the follow-up visit.
9. Subjects with a positive drug screen for illegal drugs including cannabis at Screening or Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-emergent Adverse Events | Baseline up to Follow Up/End of Treatment visit, an average of 8 months.
  Incidence and severity of adverse events, including serious adverse events and adverse events, clinically significant changes in laboratory testing, vital signs, Holter monitoring, physical examination, and ECGs
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) Response | Administered at each of the following visits in Part 3: Screening, Clinic Discharge, and Follow-up/Early Withdrawal.
  Type of Suicidal Ideation, Intensity (1 - 5, with 5 being most severe), Suicidal Behavior

SECONDARY OUTCOMES:
Pharmacokinetic Assessment | Day 1 through End of Dosing Period.
  Concentration of BMB-101 in Plasma and Urine samples:
  * SAD - 13 blood collection timepoints & 8 urine PK collection periods over 4 days (Day 1 through End of Dosing period)
  * FE - 10 blood collection timepoints over 4 days (Day 1 through End of Dosing period) - 20 blood collection timepoints in total as 2 periods in FE
  * MAD - 23 blood collection timepoints & 8 urine PK collection periods over 7 days (Day 1 through End of Dosing period)

CONTACTS AND LOCATIONS:
Overall Officials: Michele De Sciscio, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No